CLINICAL TRIAL: NCT03920722
Title: Efficacy and Safety of Rituximab in the Treatment of Good Prognosis Microscopic Polyangiitis
Acronym: RITUXGOPRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Vasculitis Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P170909J; 2018-000637-12 (EudraCT Number)
Record Dates: First submitted 2019-02-18; First posted 2019-04-19 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Microscopic Polyangiitis (MPA)
Keywords: MPA; Rituximab; ANCA-associated vasculitis
MeSH Terms: conditions — Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental): Experimental regimen: One year Glucocorticoid treatment and Rituximab IV 1 gram on Day 1 and 15
  Interventions: Drug: Rituximab
- Rituximab-Placebo (Placebo Comparator): Standard regimen: One-year Glucocorticoid treatment and Placebo-Rituximab IV on Day 1 and 15
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rituximab — 1 gram IV on Day 1 and 15 after premedication with 100 mg méthylprednisolone, 1 gramm paracetamol and 5 mg dexchlorpheniramine
  Arms: Rituximab
Drug: placebo — Placebo-Rituximab 1 gram IV on Day 1 and 15 after premedication with 100 mg méthylprednisolone, 1 gramm paracetamol and 5 mg dexchlorpheniramine
  Arms: Rituximab-Placebo

SUMMARY:
The purpose of the study is to determine wether a rituximab-based treatment compared to standard therapy (glucocorticoid alone) in patients with microscopic polyangiitis without any bad prognosis marker increases the remission and reduces the relapse free survival rate.

DETAILED DESCRIPTION:
Microscopic polyangiitis (MPA), is a small-sized vessel necrotizing vasculitis associated with anti-neutrophils cytoplasmic antibody (ANCA). Treatment of ANCA associated vasculitis (AAV) was previously based on glucocorticoids (GC) and cyclophosphamide. It has been demonstrated in two prospective randomized trials that rituximab is as effective as cyclophosphamide in the induction treatment of GPA and severe MPA. In addition, it was shown in GPA and MPA that rituximab is superior to azathioprine as maintenance therapy.

Patients with MPA without poor prognosis factor (Five factor score (FFS)=0) have not been included in the previous studies and GC alone is considered as the reference treatment in these patients. However, as much as 50% of these patients experience relapses after a 24 months follow-up and only 40% of patients have a long lasting remission.

In the group of patients with MPA without any poor prognosis factor (FFS=0), an additional treatment with rituximab might decrease the relapse rate from 40% to 15% after an 18 months' follow-up. The efficacy and safety of this proposal must be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (male or female) over 18 year old
2. Patient agree to participate in the study and signed written informed consent
3. Patient with MPA according to the CHCC established in 2012
4. Absence of any poor prognosis factor (modified five factor score (FFS) 1996 = 0)
5. Patient with recent onset or relapse of the disease (<1 month) defined by BVAS > 0, who did not received any other treatment than glucocorticoids during last month. For patients with a BVAS<3, activity of vasculitis (either relapse or new onset) has to be confirmed by the coordinating investigator. One to 3 initial glucocorticoids pulse(s) are allowed.
6. Patient with anti-MPO antibody measured by enzyme - linked immunosorbent assay (ELISA).
7. Negative pregnancy test (serum β-hCG) for women of child-bearing potential and a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study and 12 months after stopping therapy

Exclusion Criteria:

1. Small-sized vessels vasculitis not associated to anti-MPO antibody or associated with anti-PR3 positivity.
2. Patients with either GPA or EGPA vasculitis according to ACR criteria
3. Patient with a modified FFS 1996 ≥ 1
4. Patient with alveolar hemorrhage requiring mechanical ventilation
5. Patient with previous glucocorticoids treatment >1 month and > 10mg/day either for vasculitis or for any other reason.
6. Patient already receiving immunosuppressant or biological agent.

   Prior treatment with any of the following:
   * azathioprine, methotrexate, mycophenolate mophetil, mycophenolic acid within 4 weeks before inclusion
   * alkylant agent such as cyclophosphamide within 6 months before inclusion
   * anti-TNF inhibitors : infliximab within 8 weeks, adalimumab and etanercept within 2 weeks before inclusion
   * anti-CD20 therapy within one year before inclusion.
7. Patient with a previous diagnosis of cancer < 5 years (except for in situ cervical cancer and skin carcinoma with R0 resection)
8. Patient with acute infections or chronic active infections (HIV, hepatitis B or C)
9. Breast feeding woman or woman refusing the use of a contraceptive method for the 18 months' duration of the study
10. Contraindication to treatment (glucocorticoids or rituximab)
11. Unable to receive written informed consent of patient. Patient unable to understand the protocol
12. Patient already in another therapeutic protocol
13. Patient without social security
14. Patient with severe cardiac failure defined as class IV in New York Heart Association classification or severe, uncontrolled cardiac disease.
15. Patients with hypersensitivity to a monoclonal antibody or biological agent.
16. Patients in a severely immunocompromised state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-10-24 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Disease free survival rate | 18 months
  Failure free survival in patients with microscopic polyangiitis treated with rituximab and glucocorticoids compared to glucocorticoids alone.
  * Primary failure: Vasculitis requiring a modification of immunosuppressive treatment or prednisone tapering protocol before M3
  * Remission is defined by the absence of sign attributable to vasculitis and a Birmingham Vasculitis Activity Score (BVAS)=0 at M3
  * Relapse is defined after visit M3 by a BVAS>0 or the impossibility to decrease glucocorticoids according to the predefined protocol. Therefore, patients who experience a primary failure or fail to enter remission or relapse will be considered as treatment failure. Death will also be considered as a treatment failure

SECONDARY OUTCOMES:
Cumulative dose of GC in each group | 18 months
  GC dose will be recorded at each visit
Proportion of patients who achieve a complete remission defined by the absence of sign attributable to vasculitis and a BVAS=0 | 1 month
  Absence of sign attributable to vasculitis and a BVAS=0 at M3
Compare proportion of patients who relapse and time to first relapse | 18 months
  Relapse is defined after visit M3 by the reoccurrence of signs or symptoms attributable to vasculitis and a BVAS≥1 or the impossibility to decrease GC therapy according to the predefined protocol
Among patients who relapse, proportion of major relapses | 18 months
  Major relapse is defined by reappearance or worsening of disease with a BVAS≥1 and involvement of at least one major organ, a life-threatening manifestation, or both
Among patients who relapse, proportion of minor relapses | 18 months
  Minor relapse is defined by reappearance or worsening of disease with a BVAS≥1, not corresponding to a major relapse
Mortality rate | 18 months
  Proportion will be compared between groups
Quality of life:Short Form Health Survey Questionnaire (SF-36) | 18 months
  Assessed by mean variation of the SF-36 The 36-Item Short Form Health Survey questionnaire (SF-36) questionnaire includes 36 items related to eight health component (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health.) A scale has been established for each component and results vary from 0 (bad health perception) to 100 (good health perception).
Disability | 18 months
  Assessed by the mean variation of the Health Assessment Questionnaire (HAQ) Health Assessment Questionnaire (HAQ) is a questionnaire that evaluates the disability of the patient. Results vary from 0 (no assistance is needed) to 3 (patient usually needs both a special device and help from another person).
Disability | 18 months
  Assessed by the mean variation of the Euroqol 5D (EQ-5D). The EuroQol-5 dimension (EQ-5D-3L) is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D is made up of five dimensions (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression), each of which can be rated at one of three levels (no problem, some problems, extreme/severe problems). The EuroQol questionnaire also contains a visual analogue scale (EQ-VAS), where patients are asked to rate their current health state on a 0 (worst imaginable health state) to 100 (best imaginable health state) scale.
Severity of sequels linked to vasculitis as | 18 months
  Assessed by comparison of the VDI score. The Vascular Damage index score documents any organ damage that has occurred in patients since the onset of vasculitis. The score includes 64 items that are categorized into 11 groups (by organ system) and result is the summ of each damaged items.
Proportion of patients who still receive GC at the end of follow-up | 18 months
  Proportion will be compared between groups
Number and severity of side effect. | 18 months
  Record of adverse events and serious adverse events related to vasculitis or treatment in each group. Classification is made according to the CTCAE toxicity grading system.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mouthon, MD PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guillevin L, Pagnoux C, Karras A, Khouatra C, Aumaitre O, Cohen P, Maurier F, Decaux O, Ninet J, Gobert P, Quemeneur T, Blanchard-Delaunay C, Godmer P, Puechal X, Carron PL, Hatron PY, Limal N, Hamidou M, Ducret M, Daugas E, Papo T, Bonnotte B, Mahr A, Ravaud P, Mouthon L; French Vasculitis Study Group. Rituximab versus azathioprine for maintenance in ANCA-associated vasculitis. N Engl J Med. 2014 Nov 6;371(19):1771-80. doi: 10.1056/NEJMoa1404231. PMID 25372085
- [Background] Specks U, Merkel PA, Seo P, Spiera R, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Fessler BJ, Ding L, Viviano L, Tchao NK, Phippard DJ, Asare AL, Lim N, Ikle D, Jepson B, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh K, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Mueller M, Sejismundo LP, Mieras K, Stone JH; RAVE-ITN Research Group. Efficacy of remission-induction regimens for ANCA-associated vasculitis. N Engl J Med. 2013 Aug 1;369(5):417-27. doi: 10.1056/NEJMoa1213277. PMID 23902481
- [Background] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199
- [Background] Jones RB, Tervaert JW, Hauser T, Luqmani R, Morgan MD, Peh CA, Savage CO, Segelmark M, Tesar V, van Paassen P, Walsh D, Walsh M, Westman K, Jayne DR; European Vasculitis Study Group. Rituximab versus cyclophosphamide in ANCA-associated renal vasculitis. N Engl J Med. 2010 Jul 15;363(3):211-20. doi: 10.1056/NEJMoa0909169. PMID 20647198
- [Background] Samson M, Puechal X, Devilliers H, Ribi C, Cohen P, Bienvenu B, Ruivard M, Terrier B, Pagnoux C, Mouthon L, Guillevin L; French Vasculitis Study Group (FVSG). Long-term follow-up of a randomized trial on 118 patients with polyarteritis nodosa or microscopic polyangiitis without poor-prognosis factors. Autoimmun Rev. 2014 Feb;13(2):197-205. doi: 10.1016/j.autrev.2013.10.001. Epub 2013 Oct 23. PMID 24161361